CLINICAL TRIAL: NCT05238896
Title: BARIcitinib Cognitive Emotional and Neural signaTuRE (BARICENTRE)
Brief Title: BARIcitinib Cognitive Emotional and Neural signaTuRE
Acronym: BARICENTRE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties of inclusion in the study following expiry of the experimental treatment. The time required to supply the study treatment is too long to obtain conclusive results at the end of the study.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP190353; 2020-005773-27 (EudraCT Number)
Record Dates: First submitted 2022-01-04; First posted 2022-02-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Active rheumatoid arthritis; Baricitinib treatment; Mood-improving effects; MRI
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental): Patients receiving baricitinib 4mg/day for 7 days, then open label study until day 42 with all patients receiving baricitinib during 5 weeks. 20 patients in this arm will have a MRI at day 0 and day 8
  Interventions: Drug: Baricitinib Oral Tablet [Olumiant]
- Placebo (Placebo Comparator): Patients receiving placebo 4mg/day for 7 days, then open label study until day 42 with all patients receiving baricitinib during 5 weeks. 20 patients in this arm will have a MRI at day 0 and day 8
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib Oral Tablet [Olumiant] — Baricitinib 4 mg/d oral route for 42 days
  Other Names: Baricitinib
  Arms: Baricitinib
Drug: Placebo — Placebo, 4 mg/d, oral route for 7 days, then Baricitinib 4 mg/d oral route for 5 weeks
  Arms: Placebo

SUMMARY:
Rheumatoid arthritis (RA) is a frequent and disabling disease, requiring early management to achieve clinical remission. Recently, baricitinib (jak1-jak2 inhibitor) has been shown to as an efficient treatment in placebo-controlled trials, and compared to the reference treatment with TNF inhibitor (adalimumab). Its efficacy has been reported on the inflammatory parameters, but more importantly on patient-reported outcomes. Baricitinib is thought to have anti-inflammatory effects, via its inhibition of the JAK pathway. Importantly, it has also been suggested to affect mood and pain.

Hypotheses: Inhibition of JAK Kinase pathway in patients with RA will improve emotional and cognitive processing involved in mood disorders and decrease pain sensitization.

The primary objective of this study is to evaluate early emotional impact of the JAK 1/2 inhibitor Baricitinib assessed by a facial emotion recognition task. This precocious effect on emotion processing is a surrogate marker of clinical imporvement in mood.

Phase 4 study, Double-blind randomized control study with patients receiving placebo or baricitinib for 7 days, then open label study until day 42 with all patients receiving baricitinib during 5 weeks.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a frequent and disabling disease, requiring early management to achieve clinical remission. Recently, baricitinib (jak1-jak2 inhibitor) has demonstrated its efficacy compared to placebo, and compared to the reference treatment with TNF inhibitor (adalimumab). Its efficacy has been reported on the inflammatory parameters but more importantly on patient reported outcomes. Inhibition of JAK pathway could have anti-inflammatory activity but also direct action on mood and pain.

Hypotheses: Inhibition of JAK Kinase pathway in patients with RA will improve emotional and cognitive processing involved in mood disorders and decrease pain sensitization.

The primary objective of this study is to evaluate early emotional impact of the JAK 1/2 inhibitor Baricitinib assessed by Harmer's cognitive and emotional battery, This emotional aspect is a surrogate marker of future mood impact.

The primary outcome is the number of accurate responses in facial emotion recognition task at day 1 using Harmer's cognitive battery (based on Harmer & Cowen evaluation protocol at day 1).

Phase 4 study,Double-blind randomized control study with patients receiving placebo or baricitinib for 7 days, then open label study until day 42 with all patients receiving baricitinib during 5 weeks. At baseline (day 0), RA activity, mood symptoms, the number of accurate responses in facial emotion recognition task (Harmer's cognitive battery), clinical pain sensitization, will be assessed.3 follow-up research visits will be conducted at day 1, 8 and 42 (final visit) at the Pitié Salpêtrière hospital.The first intake of the Investigational medicinal product (IMP) (baricitinib or placebo) is at day 1. At day 1, the number of accurate responses in facial emotion recognition task and RA activity will be evaluated (2 to 4 hours after intake of baricitinib). At day 8 and 42, RA activity and flares, mood symptoms, the number of accurate responses in facial emotion recognition task (Harmer's cognitive battery), clinical pain sensitization, will be assessed. In each group (placebo vs Baricitinib), 20 patients will underwent a non-contrast MRI at day 0 and 8 (with evaluation of mood modification using BOLD signal during the different experimental conditions of the Cyberball task with comparison to baseline condition, and pain evaluation using fMRI-based neurological pain signature provided by Wager et al.) During the follow-up until day 42, patients will conduct questionnaires (day 15 and 29) at home about RA activity, pain (Patient pain VAS, Patient global assessment of the disease, Flare RA questionnaire) and psychometric questionnaire (Hospital Anxiety and Depression Scale)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* Diagnosis of RA according to the ACR/EULAR 2010 classification criteria
* Active rheumatoid arthritis at inclusion (defined by a Disease Activity Score (DAS28) > 3.2)
* Patient eligible for baricitinib treatment in agreement with European label and French recommendations for RA treatment with dosage of 4mg (patients with 2mg dosage will not be included to ensure patient homogeneity)
* Informed and signed consent
* Affiliation to a french social security system (beneficiary or legal)
* For child-bearing aged women, efficient contraception

Exclusion Criteria:

* Patient under tutorship or guardianship, and incapable to give informed consent
* Diagnosis of a systemic autoimmune disease other than RA
* Treatment not allowed:

  * DMARDS other than Methotrexate or Leflunomide or Hydroxychloroquine or Salazopyrine.
  * Psychotropic treatments (antidepressive drugs, benzodiazepine, mood stabilizer) during the study or the month prior the study that could change the mood evaluation.
* Laboratory exclusions: o Total white blood cell count (WBC) less than 3 x 109 cells/L o Absolute lymphocyte count (ALC) less than 0.5 x 109 cells/L o Absolute neutrophil count (ANC) less than 1 x 109 cells/L o Hemoglobin less than 8.0 g/dl o eGFR < 60 mL/min/1.73 m² based on the most recent serum creatinine (Cockroft-Gault method) o ALT or AST > 5 times upper limit of normal o Any abnormality on screening laboratory tests that, in the opinion of the investigator, could represent a risk when participating in this protocol
* Any contraindications to baricitinib treatment or to Non-contrast MRI exam
* Hypersensitivity to the active substance or to any of the excipients
* History of active tuberculosis without treatment or chronic infectious diseasewith a need of regular use of antibiotic
* Active or prior bacterial or viral infection that required treatment with antibiotics within 30 days prior to screening
* History of lymphoma or leukemia or other malignancy besides non-melanoma skin cancer within 5 years
* Uncontrolled medical condition or planned major surgery during the study
* Pregnancy or breast-feeding
* Claustrophobia
* Patient unable to understand and follow recommendations or unable to perform self-evaluation
* Participation in another interventional study or being in the exclusion period at the end of a previous study.
* Patients with current suicidal intents or behaviors, Past or present depression or anxiety will be neither a criterion for inclusion nor a criterion for non-inclusion but will be collected in case report form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of accurate responses in facial emotion recognition task | Day 1
  Percentage of accurate responses in facial emotion recognition task using Harmer's cognitive battery (based on Harmer & Cowen evaluation protocol)

SECONDARY OUTCOMES:
DIfference in disease activity | Day 0, 8 and 42
  DIfference in disease activity on DAS28 (disease activity score on 28 joints) - SDAI (Simplified Disease Activity Score)
Difference in function improvement | Day 0, 8 and 42
  Difference in function improvement on HAQ (health assessment questionnaire)
Difference in pain | Day 0, 8 and 42
  Difference in pain using Visual Analogic Scale (VAS) for pain
Difference in patient global assessment of the disease | Day 0, 8 and 42
  Difference in VAS for patient global assessment of the disease
Number of accurate responses in facial emotion recognition task | Day 8
  The number of accurate responses in facial emotion recognition task using Harmer's cognitive battery (based on Harmer & Cowen evaluation protocol)
Difference in central and peripheral pain sensitization | Day 0, 8 and 42
  Difference in central and peripheral pain sensitization using quantitative sensory testing
Difference in the results of psychometric questionnaire | Day 0, 8 and 42
  Difference in the results of psychometric questionnaire using Hospital Anxiety and Depression Scale
Difference in blood-oxygen-level dependent (BOLD) signal activity in regions of interest (ROI) such as the subgenual anterior cingulate cortex (Sg-ACC) during a cyberball task | day 0 and day 8
  Main effect of group on social exclusion-related brain responses (e.g. actiavtion of the Sg_ACC ROI)
Difference in BOLD signal activity in pain-encoding brain regions | day 0 and day 8
  Main effect of group in pain-related brain responses
Differences in mood and pain assessments between patients with high or low expectations of the drug | Day 1,8 and 42
  Main effect of group on accurate responses during the facial emotion recognition task and pain assessment variables
Difference in BOLD signal activity in reward-learning related brain regions | day 0 and day 8
  Main effect of group reward-learning related brain responses (e.g. activation of the ventral striatum or vmPFC ROIs)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FAUTREL, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Florian BAILLY, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodological sound proposal.